CLINICAL TRIAL: NCT04814446
Title: Efficacy of the Nonavalent HPV Vaccine in the Treatment of Difficult-to-treat Palmo-plantar Warts
Brief Title: Nonavalent HPV Vaccine in the Treatment of Difficult-to-treat Palmo-plantar Warts
Acronym: VAC-WARTS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APHP200046; 2024-513671-40-00 (EU CTIS Number)
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-01

CONDITIONS: Palmar or Plantar Warts
Keywords: WARTS; Vaccine HPV
MeSH Terms: conditions — Warts | interventions — Vaccination

STUDY DESIGN:
Intervention Model Description: Multicenter national clinical trial, phase III, two parallel group randomized (in a 1:1 ratio)
Who Masked: Participant, Investigator
Masking Description: Double blind clinical trial.The identity of Gardasil 9® vaccine and placebo cannot be concealed as presentation. They will be packed in boxes of identical appearance to achieve double blindness. During the study designated unblinded trained and qualified site staff will be responsible for preparing the Gardasil 9® vaccine or placebo out of view of patients and an unblinded nurse(s) or physician(s) will be responsible for administering the study products to the patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gardasil 9® (Experimental): Nonavalent HPV vaccine
  Interventions: Biological: Vaccination
- Placebo (Placebo Comparator): NaCl 0.9 % solution for injection
  Interventions: Biological: Vaccination

INTERVENTIONS:
Biological: Vaccination — Intramuscular injections of 0,5 ml will be administered at M0, M2 and M6

SUMMARY:
Cutaneous viral warts are very common and are caused by the human papilloma virus (HPV). Most people experience warts in one form or another at some point in their lives. Cutaneous warts are related to different types of HPV. For the palms and soles, HPV 2 has been the most frequently found but HPV 1, 4, 27, and 57 have also been described. Our hypothesis is that vaccination by nonavalent vaccine against HPV could lead to a complete resolution of difficult-to-treat palmo-plantar warts patients of more than 15 years and 3 months of age.

DETAILED DESCRIPTION:
The qHPV and nHPV has been used as a therapeutic approached for the treatment of cutaneous warts in case reports and some case series. Very recently, the Journal of the American Academy of Dermatology (JAAD)-the journal with the highest impact factor in the dermatological field- has published a review of all the cases reported in the scientific literature. The authors were strongly in favor of the use of the vaccine in case of difficult-to-treat warts and have highlighted the need for clinical trials. In the literature, 80 patients have been described with cutaneous warts treated by qHPV or nHPV with more than 50% of efficacy.Our hypothesis is that vaccination by nonavalent vaccine against HPV could lead to a complete resolution of difficult-to-treat palmo-plantar warts patients of more than 15 years and 3 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Patients of age ≥ 15 years and 3 months with palmar or plantar warts (including periungueal and back of hands or feet warts) since more than one year with:
* ≥ 5 warts (X palmar and X plantar) or
* ≥ 4 cm2 of Total surface involved by the warts (Y cm x Z cm).
* Patients should have received two lines of treatment during the past year before inclusion, the last treatment must be at 3 weeks maximum before inclusion:
* At total one month of application of topical salicylic acid, with minimum 3 weeks continuous.
* At least two sprays of liquid nitrogen (two applications at the same session, or at different sessions with a few intervals).
* Painful warts (VAS ≥ 4) or functional discomfort (Revised foot function index (RFFI) or Cochin Hand Function Scale (CHSF) or social discomfort (DLQI)).
* No topical or systemic immunosuppresive/ immunomodulating drugs
* Women of childbearing potential must have a negative pregnancy test and an effective contraception (V1) and up the end of the vaccination period of 6 months;
* Individuals affiliated to a social security regimen;
* Individuals able to participate and to follow up during the study period.

Exclusion Criteria:

* Suspicion of COVID, with confirmation by autotest.
* Any causes of immunosupression: organ transplant recipients, bone-marrow transplantation, immunosupressive regimens for any diseases, HIV positivity.
* Women or men who received HPV Vaccine previously of the study;
* Any serious chronic or progressive disease according to the judgement of the investigator;
* Individuals with history of known allergies/hypersensitivity to any component of study vaccine;
* Individuals who have any malignancy or lymphoproliferative disorder;
* Individuals with thrombocytopenia or coagulation disorder contre-indicating intramusculary injections;
* Patient with anticoagulant therapy
* Individuals with body temperature > 38.0 degrees Celsius or/and acute disease within 3 days of intended study vaccination;
* Women who are pregnant or are breast-feeding, or are of childbearing age who have not used or do not plan to use acceptable birth control measures, during the first 6 months ½ of the study;
* Individuals under a measure of legal protection or unable to consent;
* Individuals participating in any clinical trial with another investigational product 28 days prior to first study visit or intent to participate in another clinical study at any time during the conduct of the study.
* Participation in another interventional study involving human participants or being in the exclusion period at the end of a previous study involving human participants, if applicable
* Patient on AME (state medical aid) (unless exemption from affiliation).
* Patient wishing to be vaccinated with Gardasil 9® within 6 months or refusing the principle of postponing vaccination.
* Immunosuppressive therapy including use of systemic corticosteroids or chronic immunosuppressant medication (more than 14 days)

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2022-06-29 (Actual); Primary Completion 2025-06-29 (Estimated); Study Completion 2026-06-29 (Estimated)

PRIMARY OUTCOMES:
Complete remission of cutaneous warts | 7 months
  Complete remission of cutaneous warts 7 months after the first injection of the vaccine

SECONDARY OUTCOMES:
Quality of Life evaluated | Inclusion, 2 months, 6 months, 7 months
  Quality of Life will be evaluated with QoL Questionnaire (DLQI)
Pain (VAS) | Inclusion, 2 months, 6 months, 7 months
  Pain will be assess using VAS
Functional discomfort for walking and functional disability in hands | Inclusion, 2 months, 6 months, 7 months
  Functional discomfort for walking and functional disability in hands will be evaluated using the Revised Foot Function index or Cochin hand function scale respectively at M0, M2, M6, M7.
Partial remission of cutaneous warts | 7 months
  Partial remission of cutaneous warts 7 months after the first injection of the vaccine.
Number of warts appeared | Inclusion, 2 months, 6 months, 7 months
  Number of warts appeared at M2, M6, M7

CONTACTS AND LOCATIONS:
Overall Officials: Johan CHANAL, Dr, Principal Investigator — Hospital Cochin; Olivier CHOSIDOW, Pr, Study Director — Henri Mondor University Hospital
Locations (1):
- Hospital Cochin, Paris, France

IPD SHARING:
Plan to Share IPD: No